CLINICAL TRIAL: NCT01718535
Title: Method Comparison Study of the Spartan FRX CYP2C19 *2, *3, and *17 Genotyping System
Brief Title: Method Comparison Study of the Spartan FRX CYP2C19 Genotyping System Against Bi-directional Sequencing
Status: Completed | Type: Observational
Sponsor: Spartan Bioscience Inc. (Industry)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 01001679
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-05

CONDITIONS: Genotyping Techniques
Keywords: Cyp2C19; Genotyping; Spartan; Comparison; Sequencing

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CYP2C19 Genotyping
  Interventions: Device: Spartan FRX CYP2C19 Test System

INTERVENTIONS:
Device: Spartan FRX CYP2C19 Test System

SUMMARY:
The Spartan FRX CYP2C19 Test System (hereafter referred to as the 'FRX System') is a qualitative in vitro diagnostic test for the identification of a patient's CYP2C19 *2, *3 and *17 genotypes from genomic DNA obtained from buccal swab samples. This study is purposed to demonstrate the concordance (positive and negative percent agreement) by comparing the Spartan FRX system against bi-directional DNA sequencing. The study will also evaluate the concordance between three different sample transport embodiments provided to laboratories for use in transporting the reagent tubes with collected buccal sample swab to the laboratory.

DETAILED DESCRIPTION:
The Spartan FRX CYP2C19 Test System (hereafter referred to as the 'FRX System') is a qualitative in vitro diagnostic test for the identification of a patient's CYP2C19 *2, *3 and *17 genotypes from genomic DNA obtained from buccal swab samples.

The FRX system is comprised of hardware and consumable components. The hardware components of the system include an Analyzer (thermal cycler with fluorescence detection capability), a netbook computer and a printer. The consumable component of the FRX system is a sample collection kit. Each kit contains a buccal swab (used to collect the patient sample) and a tube containing the reagents required for genomic DNA extraction and PCR amplification stages of the test.

The Spartan FRX System is capable of detecting three CYP2C19 SNPs (*2, *3, *17) in each test performed. An individual sample collection kit is required for each SNP tested; therefore three sample collection kits are required for each test performed on the system.

The FRX System is to be used by trained personnel in CLIA certified laboratories and is for use with buccal samples collected directly from patients. The FRX CYP2C19 test is intended to enable clinicians to identify patients with mutations in the *2,*3 and *17 loci of the CYP2C19 gene and is indicated for use as an aid to clinicians in determining strategies for therapeutics that are metabolized by the CYP2C19 gene product.

To perform a test, the user collects three buccal samples from the patient and then inserts a sample into each of the three reagent tubes (one for each of the CYP2C19 loci *2, *3 and *17). The reagent tubes are placed into the Analyzer and the FRX system automates the processes of DNA extraction, PCR amplification, fluorescent signal detection and data analysis. The system provides the user with a printed result listing the patient genotypes at the *2, *3 and *17 loci.

This study has been designed to demonstrate the concordance (positive and negative percent agreement) by comparing the Spartan FRX system against bi-directional DNA sequencing. The study will also evaluate the concordance between three different sample transport embodiments provided to laboratories for use in transporting the reagent tubes with collected buccal sample swab to the laboratory.

For each mutation, agreement of the FRX System against bidirectional sequencing (comparative method) will be calculated: The overall accuracy of the test will be calculated and reported as follows:

* of concordant results between the test and the reference method Accuracy = ----------------------------------------------------------------
* of samples analyzed by the reference method

The first and second pass results from the study will be analyzed and tabulated as outlined in the table below. The acceptance criteria for the overall study will be percent in agreement ≥ 99.0% for the second pass with the lower bound of a one-sided 95% confidence interval using the score method ≥ 95.0%.

ELIGIBILITY:
Exclusion Criteria:

None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 320 Individuals with undetermined CYP2C19 *2 *3 and *17 Genotypes
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azar Azad, PhD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Services, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of study participants was performed without knowledge of participant genotypes by enrolling associates of operators and associates of Spartan Bioscience and Mount Sinai Services.
Period: Overall Study
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *1/*3 CYP2C19 Genotype | *3/*3 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype | *3/*17 CYP2C19 Genotype
Started | 131 | 95 | 19 | 8 | 1 | 40 | 11 | 6 | 15 | 1
First Pass | 128 | 94 | 19 | 7 | 1 | 39 | 11 | 6 | 15 | 1
Completed | 130 | 95 | 19 | 7 | 1 | 40 | 11 | 6 | 15 | 1
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Bidirectional Sequencing not possible | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *1/*3 CYP2C19 Genotype | *3/*3 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype | *3/*17 CYP2C19 Genotype | Total
Number analyzed (Participants) | 130 | 95 | 19 | 7 | 1 | 40 | 11 | 6 | 15 | 1 | 325
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5
  Between 18 and 65 years | 124 | 95 | 19 | 7 | 1 | 38 | 9 | 6 | 15 | 1 | 315
  >=65 years | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5
Sex/Gender, Customized [Number; unit: Participants]
  Gender Not Collected | 130 | 95 | 19 | 7 | 1 | 40 | 11 | 6 | 15 | 1 | 325
Region of Enrollment [Number; unit: participants]
  Canada | 130 | 95 | 19 | 7 | 1 | 40 | 11 | 6 | 15 | 1 | 325

OUTCOME MEASURES:

1. Primary Outcome: Percent Agreement
Description: The study will pass if the percent agreement is ≥ 99.0% and the lower bound of a 1-sided 95% confidence interval is ≥ 95.0% using the score method.
Time Frame: After second pass result is complete (~3hours)
Measure: Number (95% Confidence Interval); unit: Percent Agreement
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *1/*3 CYP2C19 Genotype | *3/*3 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype | *3/*17 CYP2C19 Genotype
Number analyzed (Participants) | 130 | 95 | 19 | 7 | 1 | 40 | 11 | 6 | 15 | 1
Percent Agreement | 100 [98 to 100] | 100 [97 to 100] | 100 [88 to 100] | 100 [72 to 100] | 100 [27 to 100] | 100 [94 to 100] | 100 [80 to 100] | 100 [69 to 100] | 100 [85 to 100] | 100 [27 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the full duration of the trial (~1 months).
Description: No adverse events were encountered.
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *1/*3 CYP2C19 Genotype | *3/*3 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype | *3/*17 CYP2C19 Genotype
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/95 | 0/19 | 0/8 | 0/1 | 0/40 | 0/11 | 0/6 | 0/15 | 0/1
Other Adverse Events (participants affected / at risk) | 0/131 | 0/95 | 0/19 | 0/8 | 0/1 | 0/40 | 0/11 | 0/6 | 0/15 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less